CLINICAL TRIAL: NCT06553404
Title: A Prospective, Randomized, Controlled Double Masked Trial to Assess the Performance of Myoslow Lens in Slowing Myopia Progression in Children
Brief Title: Myoslow Lens Study to Control Myopia in Children
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Crystal Optic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLD-001
Record Dates: First submitted 2024-07-28; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and site staff will be masked to the assigned arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single vision (Active Comparator): Single vision glasses
  Interventions: Device: Single Vision
- myoslow (Experimental): The Myoslow spectacle lens is based on the Defocus Incorporated Multiple Segments (DIMS) mechanism of action. This lens provides the same optical image as the Defocusing Incorporated Soft Contact Lens (DISC) without the drawbacks inherent with contact lens fitting.
  Interventions: Device: Myoslow

INTERVENTIONS:
Device: Myoslow — The Myoslow spectacle lens is based on the Defocus Incorporated Multiple Segments (DIMS) mechanism of action. This lens provides the same optical image as the Defocusing Incorporated Soft Contact Lens (DISC) without the drawbacks inherent with contact lens fitting.
  Arms: myoslow
Device: Single Vision — Single vision glasses
  Arms: Single vision

SUMMARY:
A Prospective, randomized, controlled double masked trial to assess the performance of Myoslow lens in slowing myopia progression in children.

The following study measures will be assessed:

* Demographics and medical history
* Current spectacles
* Best Corrected Visual Acuity (BCVA) assessed by Measurement and Summation (M&S) system
* Biometry
* Cover test
* Stereopsis
* Ocular Motility
* Pupil responses
* Cycloplegic refraction
* Fundus Examination
* Vision related quality of life using the questionnaire Pediatric Refractive Error Profile (PREP)2
* Adverse Events

ELIGIBILITY:
Inclusion Criteria:

* Children, 6-12 years old
* Spherical Equivalence Refraction (SER): -1.00 to -5.00 Diopter (D).
* Astigmatism and anisometropia of 1.50 D or less.
* Best Corrected Visual Acuity (BCVA) (6 / 7.5) or higher.

Exclusion Criteria:

* Eye and systemic disorders.
* Previously treated for myopia

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
spherical equivalent error | 24 months
  Change in spherical equivalent refractive error from baseline to 24-month visit

SECONDARY OUTCOMES:
Axial length | 24 months
  Mean change in axial length (mm) from baseline at 24-month visit (Based on Biometry)

CONTACTS AND LOCATIONS:
Overall Officials: Haim Stolovitch, MD, Study Chair — Crystal Optic
Locations (1):
- Sheba MC, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No
coded data only